CLINICAL TRIAL: NCT03432520
Title: A Multi-Center Evaluation of the Long-Term Safety and Efficacy of Spark-sponsored Gene Therapies in Males With Hemophilia A
Brief Title: Long-Term Safety and Efficacy of Spark-Sponsored Gene Therapies in Males With Hemophilia A
Status: Active, not recruiting | Type: Observational
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPK-8011/8016-LTFU
Record Dates: First submitted 2018-01-24; First posted 2018-02-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Genetic: SPK-8011 — Observational long-term safety follow-up study of participants previously treated with SPK-8011 in any Spark-sponsored SPK-8011 study
Genetic: SPK-8016 — Observational long-term safety follow-up study of participants previously treated with SPK-8016 in any Spark-sponsored SPK-8016 study

SUMMARY:
This long-term follow-up study will continue to evaluate the long-term safety and efficacy of SPK-8011 and SPK-8016 in males with hemophilia A, who have received a single intravenous administration of SPK-8011 or SPK-8016 in any Spark-sponsored SPK-8011 or SPK-8016 study.

DETAILED DESCRIPTION:
This study will follow patients with hemophilia A, who have received a single intravenous administration of SPK-8011 or SPK-8016 in any prior Spark-sponsored SPK-8011 or SPK-8016 study. Participants will be followed for up to a total of 10 years post infusion (including the time on the dosing study).

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Have received a single intravenous administration of SPK-8011 or SPK-8016 in either Study SPK-8011-101 or SPK-8016-101, respectively.
2. Understand the purpose and risks of the study and provide signed and dated informed consent before undergoing any study-specific procedures.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1.Unable or unwilling to comply with the schedule of visits and study assessments as described in this study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetic males
Study Population: Males with hemophilia A, who received a single intravenous administration of SPK-8011 or SPK-8016 in any Spark-sponsored study.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 9 years
Number of Participants with Adverse Events of Special Interest (AESIs) | Up to 9 years
Incidence of Coagulation Factor VIII (FVIII) Inhibitor Development | Up to 9 years
Number of Participants with Clinical Laboratory Abnormalities | Up to 9 years
Number of Participants with Vital Sign Abnormalities | Up to 9 years
Number of Participants with Physical Exam Abnormalities | Up to 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Director, Study Director — Spark Therapeutics, Inc.
Locations (12):
- United States (9):
  - Boston Children's Hospital, Boston, Massachusetts
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Truman Medical Centers, Kansas City, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Pennsylvania State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Royal Prince Alfred Hospital Department of Cell & Molecular Therapies, Sydney, New South Wales
  - The Alfred Hospital & Monash Medical Centre, Melbourne, Victoria
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] George LA, Monahan PE, Eyster ME, Sullivan SK, Ragni MV, Croteau SE, Rasko JEJ, Recht M, Samelson-Jones BJ, MacDougall A, Jaworski K, Noble R, Curran M, Kuranda K, Mingozzi F, Chang T, Reape KZ, Anguela XM, High KA. Multiyear Factor VIII Expression after AAV Gene Transfer for Hemophilia A. N Engl J Med. 2021 Nov 18;385(21):1961-1973. doi: 10.1056/NEJMoa2104205. PMID 34788507